CLINICAL TRIAL: NCT03137446
Title: Assessing Targeted Fluid Resuscitation Strategies Among Patients With Severe Sepsis and Septic Shock
Brief Title: Restrictive Intravenous Fluids Trial in Sepsis
Acronym: RIFTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 409916
Record Dates: First submitted 2017-04-10; First posted 2017-05-02 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-06

CONDITIONS: Septic Shock; Severe Sepsis
Keywords: Intravenous fluid resuscitation; Septic shock; Severe sepsis; Fluid restriction
MeSH Terms: conditions — Shock, Septic; Sepsis

STUDY DESIGN:
Intervention Model Description: Randomized Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Participants randomized to the usual care resuscitation strategy will receive an initial 30 ml/kg bolus and then IV fluids as needed and without limit as well as IV vasopressors to maintain a MAP>65, determined by the primary care team for the duration of the study.
- Restrictive Care (Experimental): Participants randomized to the restrictive fluid resuscitation strategy will be LIMITED to 60 ml/kg (up to 6000 ml) of IV fluids as initial resuscitation followed by administration of IV vasopressors to maintain a MAP>65 mm Hg for the first 72 hours of care. The intervention is defined as capping the total allowed IVF administered. After 72 hours the participants are eligible for IV fluids as determined by the primary care team.
  Interventions: Other: Intravenous Fluid Cap

INTERVENTIONS:
Other: Intravenous Fluid Cap — Normal Saline or Ringers Lactate limited to 60ml/kg for first 72 hours
  Arms: Restrictive Care

SUMMARY:
IV fluid resuscitation has long been recognized to be an important treatment for patients with severe sepsis and septic shock. While under-resuscitation is known to increase morbidity and mortality, contemporary data suggests that overly aggressive fluid resuscitation may also be harmful. Currently, following an initial IVF resuscitation of 30 ml/kg, there is no standard of care and a lack of evidence to support a fluid restrictive or more liberal strategy. The investigators seek to determine if a fluid restrictive strategy reduces morbidity and mortality among patients with severe sepsis and septic shock.

DETAILED DESCRIPTION:
Sepsis is one of the most common indications for intensive care unit admission world wide and the third leading cause of death in the United States. While IV fluid administration has been recognized as an important part of sepsis resuscitation for over 15 years, there is growing concern that overly aggressive IV fluid resuscitation may be harmful to patients with severe sepsis and septic shock.

The current standard of care for initial resuscitation is outlined in the 2016 Surviving Sepsis guidelines which recommends a 30mL/kg bolus of IV fluid for septic patients with hypotension (mean arterial pressure <65 mm Hg) or a lactic acid >4mmol/L within the first 3 hours of presentation. This standard is affirmed by the 2015 Centers for Medicare & Medicaid (CMS) SEP-1 guidelines. Afterwards, the guidelines advise the use of vasopressors to maintain a mean arterial pressure (MAP) of >65 mm Hg within the first 6 hours of patient care. Following the initial 30mL/kg bolus, there is no established standard of care for fluid administration; therefore there is significant variation in care between providers and institutions. Currently, there is no human data that indicates that larger volume (>30mL/kg) resuscitation strategy improves blood pressure or end organ perfusion , yet it is not uncommon for patients to receive large volumes of IV fluid (5-10 liters) in the early stages of resuscitation.

When considering how much IV fluids are typically administered to patients with septic shock, examination of the large EGDT RCTs provides a more informed picture. In the original Rivers study patients received approximately 70 mL/kg of IVF in the first 6 hours and additional 125 ml/kg in hours 7 to 72.3 Notably, this large volume resuscitation did not produce increased rates of clinically important heart failure and intubation. In the contemporary EGDT validation trials, patients received 60-70 ml/kg of IVF in the first 6 hours and only 60-70 ml/kg from hours 7 to 72.6,7,8 The contemporary alternative approach being advocated among critical care practitioners is to use vasopressors to maintain a mean arterial pressures above 65 mm Hg following the initial 30 ml/kg bolus, thereby maintaining organ perfusion, while limiting further IV fluid administration.9 Without clear evidence to guide physicians under current usual care the amount of IV fluid administration varies widely between providers and institutions when resuscitating patients with severe sepsis and septic shock.

The investigators hypothesize the use of a fluid restrictive strategy will result in a lower 28-day mortality, ICU length of stay and total number of ventilator days but will not reduce the number of patients who need hemodialysis or require intubation.

The primary outcome of the study is to assess if a restrictive IV fluid resuscitation strategy has a composite benefit of a reduced discharge mortality or Persistent Organ Dysfunction (POD) score compared to a usual care among patients with severe sepsis and septic shock. POD is defined by the ongoing need for vasopressor agents such as norepinephrine, epinephrine, vasopressin or dopamine for more than two hours in a given day; persistent renal failure as defined by the need for any ongoing renal replacement therapy; and persistent respiratory/neuromuscular failure as defined by the ongoing need for mechanical ventilation (not including non-invasive ventilation modalities).

ELIGIBILITY:
Inclusion Criteria:

1. The patients must be suspected by the treating physician to have sepsis causing their acute illness as exhibited by 2 or more of the following Systemic Inflammatory Response Syndrome (SIRS) criteria was well as a known or suspected infection at the time of screening:

   1. Temperature of > 38 C or < 36 C
   2. Heart rate of > 90/min
   3. Respiratory rate of > 20/min or PaCO2 < 32 mm Hg
   4. White blood cell count > 12000/mm3 or < 4000/mm3 or >10% immature bands.
2. Since approximately 12% of patients ultimately diagnosed with sepsis do not meet SIRS criteria , SIRS negative patients will be eligible for the study if the treating physician makes a clinical diagnosis of severe sepsis or septic shock.
3. Patients must be suspected of having severe sepsis or septic shock defined as refractory hypotension or a lactic acid>4 at the time of enrollment. Refractory hypotension is defined as having a SBP <90 or MAP <65, for 15 minutes, following 1000 mL of IV fluid or a blood pressure maintained by vasopressor administration.
4. Patients must have received less than 60ml/kg of intravenous fluid at time of study enrollment.

Exclusion Criteria:

1. Patients with a PRIMARY diagnosis of acute cerebral vascular event, acute coronary syndrome, acute pulmonary edema, status asthmaticus, active gastrointestinal bleeding, seizure, drug overdose, burn, trauma, requirement for immediate surgery, or undergoing extracorporeal membrane oxygenation.
2. Patients who have a diagnosis of severe sepsis or septic shock and additionally have an active fluid wasting process such as extensive diarrhea, diabetes insipidus, cerebral salt wasting, or an osmotic diuresis.
3. Patients who have a diagnosis of severe sepsis or septic shock who have a concurrent diagnosis of diabetic ketoacidosis, hyperosmolar non-ketotic hyperglycemia, or rhabdomyolysis.
4. Patients who have received >60 ml/kg of IVF resuscitation.
5. Patient who are <18 years old, pregnant, or incarcerated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Discharge Mortality and Persistent Organ Dysfunction (POD) a composite outcome | At participant hospital discharge or up to 60 days
  Persistent Organ Dysfunction is defined as the ongoing need for vasopressor agents such as norepinephrine, epinephrine, vasopressin or dopamine for more than two hours in a given day; persistent renal failure as defined by the need for any ongoing renal replacement therapy; or persistent respiratory failure as defined by the ongoing need for mechanical ventilation at least 2 hours a day. The composite outcome will be defined as having at least one of the 4 possible composite outcomes (death, vasopressor support, persistent renal failure, or persistent respiratory failure). If a patient has one or more of these outcomes they will be classified as having the primary composite outcome. If the patient has 0 of 4 outcomes they will be classified as not having the composite outcome.

SECONDARY OUTCOMES:
7 day Mortality and Persistent Organ Dysfunction | Day 7
  Persistent Organ Dysfunction is defined as the ongoing need for vasopressor agents such as norepinephrine, epinephrine, vasopressin or dopamine for more than two hours in a given day; persistent renal failure as defined by the need for any ongoing renal replacement therapy; or persistent respiratory failure as defined by the ongoing need for mechanical ventilation at least 2 hours a day. The composite outcome will be defined as having at least one of the 4 possible composite outcomes (death, vasopressor support, persistent renal failure, or persistent respiratory failure). If a patient has one or more of these outcomes they will be classified as having the secondary composite outcome. If the patient has 0 of 4 outcomes they will be classified as not having the composite outcome.
30 day Mortality and Persistent Organ Dysfunction | Day 30
  Persistent Organ Dysfunction is defined as the ongoing need for vasopressor agents such as norepinephrine, epinephrine, vasopressin or dopamine for more than two hours in a given day; persistent renal failure as defined by the need for any ongoing renal replacement therapy; or persistent respiratory failure as defined by the ongoing need for mechanical ventilation at least 2 hours a day. The composite outcome will be defined as having at least one of the 4 possible composite outcomes (death, vasopressor support, persistent renal failure, or persistent respiratory failure). If a patient has one or more of these outcomes they will be classified as having the secondary composite outcome. If the patient has 0 of 4 outcomes they will be classified as not having the composite outcome.
60 day Mortality and Persistent Organ Dysfunction | Day 60
  Persistent Organ Dysfunction is defined as the ongoing need for vasopressor agents such as norepinephrine, epinephrine, vasopressin or dopamine for more than two hours in a given day; persistent renal failure as defined by the need for any ongoing renal replacement therapy; or persistent respiratory failure as defined by the ongoing need for mechanical ventilation at least 2 hours a day. The composite outcome will be defined as having at least one of the 4 possible composite outcomes (death, vasopressor support, persistent renal failure, or persistent respiratory failure). If a patient has one or more of these outcomes they will be classified as having the secondary composite outcome. If the patient has 0 of 4 outcomes they will be classified as not having the composite outcome.
Intensive Care Unit length of stay | up to 60 days
  Number of hours the participant spends in the ICU
Length of Shock | up to 60 days
  Number of hours of shock requiring vasopressors
Requirement for renal replacement therapy or reduction of renal failure | up to 60 days
  Need for intermittent or continuous or intermittent hemodialysis
Mechanical Intubation | up to 60 days
  Proportion of patients intubated during their ICU course
Hyperchloremic metabolic acidosis | up to 60 days
  Development of a non anion gap metabolic acidosis secondary to hyperchloremia
Time of mechanical ventilation | up to 60 days
  For those patients intubated, the number of hours that they received mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Keith Corl, MD, Principal Investigator — Department of Pulmonary Critical Care Brown University; Mitchell Levy, MD, Study Chair — Department of Pulmonary Critical Care Brown University; Amy Palmisciano, RN, BSN, Study Director — Department of Pulmonary Critical Care Brown University
Locations (1):
- Rhode Island Hosptial, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Angus DC, Linde-Zwirble WT, Lidicker J, Clermont G, Carcillo J, Pinsky MR. Epidemiology of severe sepsis in the United States: analysis of incidence, outcome, and associated costs of care. Crit Care Med. 2001 Jul;29(7):1303-10. doi: 10.1097/00003246-200107000-00002. PMID 11445675
- [Background] Vincent JL, Sakr Y, Sprung CL, Ranieri VM, Reinhart K, Gerlach H, Moreno R, Carlet J, Le Gall JR, Payen D; Sepsis Occurrence in Acutely Ill Patients Investigators. Sepsis in European intensive care units: results of the SOAP study. Crit Care Med. 2006 Feb;34(2):344-53. doi: 10.1097/01.ccm.0000194725.48928.3a. PMID 16424713
- [Background] Rivers E, Nguyen B, Havstad S, Ressler J, Muzzin A, Knoblich B, Peterson E, Tomlanovich M; Early Goal-Directed Therapy Collaborative Group. Early goal-directed therapy in the treatment of severe sepsis and septic shock. N Engl J Med. 2001 Nov 8;345(19):1368-77. doi: 10.1056/NEJMoa010307. PMID 11794169
- [Background] Holst LB, Haase N, Wetterslev J, Wernerman J, Guttormsen AB, Karlsson S, Johansson PI, Aneman A, Vang ML, Winding R, Nebrich L, Nibro HL, Rasmussen BS, Lauridsen JR, Nielsen JS, Oldner A, Pettila V, Cronhjort MB, Andersen LH, Pedersen UG, Reiter N, Wiis J, White JO, Russell L, Thornberg KJ, Hjortrup PB, Muller RG, Moller MH, Steensen M, Tjader I, Kilsand K, Odeberg-Wernerman S, Sjobo B, Bundgaard H, Thyo MA, Lodahl D, Maerkedahl R, Albeck C, Illum D, Kruse M, Winkel P, Perner A; TRISS Trial Group; Scandinavian Critical Care Trials Group. Lower versus higher hemoglobin threshold for transfusion in septic shock. N Engl J Med. 2014 Oct 9;371(15):1381-91. doi: 10.1056/NEJMoa1406617. Epub 2014 Oct 1. PMID 25270275
- [Background] Jones AE, Shapiro NI, Trzeciak S, Arnold RC, Claremont HA, Kline JA; Emergency Medicine Shock Research Network (EMShockNet) Investigators. Lactate clearance vs central venous oxygen saturation as goals of early sepsis therapy: a randomized clinical trial. JAMA. 2010 Feb 24;303(8):739-46. doi: 10.1001/jama.2010.158. PMID 20179283
- [Background] ProCESS Investigators; Yealy DM, Kellum JA, Huang DT, Barnato AE, Weissfeld LA, Pike F, Terndrup T, Wang HE, Hou PC, LoVecchio F, Filbin MR, Shapiro NI, Angus DC. A randomized trial of protocol-based care for early septic shock. N Engl J Med. 2014 May 1;370(18):1683-93. doi: 10.1056/NEJMoa1401602. Epub 2014 Mar 18. PMID 24635773
- [Background] Mouncey PR, Osborn TM, Power GS, Harrison DA, Sadique MZ, Grieve RD, Jahan R, Harvey SE, Bell D, Bion JF, Coats TJ, Singer M, Young JD, Rowan KM; ProMISe Trial Investigators. Trial of early, goal-directed resuscitation for septic shock. N Engl J Med. 2015 Apr 2;372(14):1301-11. doi: 10.1056/NEJMoa1500896. Epub 2015 Mar 17. PMID 25776532
- [Background] ARISE Investigators; ANZICS Clinical Trials Group; Peake SL, Delaney A, Bailey M, Bellomo R, Cameron PA, Cooper DJ, Higgins AM, Holdgate A, Howe BD, Webb SA, Williams P. Goal-directed resuscitation for patients with early septic shock. N Engl J Med. 2014 Oct 16;371(16):1496-506. doi: 10.1056/NEJMoa1404380. Epub 2014 Oct 1. PMID 25272316
- [Background] Marik PE. Early management of severe sepsis: concepts and controversies. Chest. 2014 Jun;145(6):1407-1418. doi: 10.1378/chest.13-2104. PMID 24889440
- [Background] Dellinger RP, Levy MM, Rhodes A, Annane D, Gerlach H, Opal SM, Sevransky JE, Sprung CL, Douglas IS, Jaeschke R, Osborn TM, Nunnally ME, Townsend SR, Reinhart K, Kleinpell RM, Angus DC, Deutschman CS, Machado FR, Rubenfeld GD, Webb S, Beale RJ, Vincent JL, Moreno R; Surviving Sepsis Campaign Guidelines Committee including The Pediatric Subgroup. Surviving Sepsis Campaign: international guidelines for management of severe sepsis and septic shock, 2012. Intensive Care Med. 2013 Feb;39(2):165-228. doi: 10.1007/s00134-012-2769-8. Epub 2013 Jan 30. PMID 23361625
- [Background] Hilton AK, Bellomo R. A critique of fluid bolus resuscitation in severe sepsis. Crit Care. 2012 Jan 25;16(1):302. doi: 10.1186/cc11154. PMID 22277834
- [Background] Hilton AK, Bellomo R. Totem and taboo: fluids in sepsis. Crit Care. 2011;15(3):164. doi: 10.1186/cc10247. Epub 2011 Jun 10. PMID 21672278
- [Background] Landry DW, Oliver JA. The pathogenesis of vasodilatory shock. N Engl J Med. 2001 Aug 23;345(8):588-95. doi: 10.1056/NEJMra002709. No abstract available. PMID 11529214
- [Background] Ueda S, Nishio K, Akai Y, Fukushima H, Ueyama T, Kawai Y, Masui K, Yoshioka A, Okuchi K. Prognostic value of increased plasma levels of brain natriuretic peptide in patients with septic shock. Shock. 2006 Aug;26(2):134-9. doi: 10.1097/01.shk.0000226266.99960.d0. PMID 16878020
- [Background] Zhang Z, Zhang Z, Xue Y, Xu X, Ni H. Prognostic value of B-type natriuretic peptide (BNP) and its potential role in guiding fluid therapy in critically ill septic patients. Scand J Trauma Resusc Emerg Med. 2012 Dec 31;20:86. doi: 10.1186/1757-7241-20-86. PMID 23276277
- [Background] Bruegger D, Jacob M, Rehm M, Loetsch M, Welsch U, Conzen P, Becker BF. Atrial natriuretic peptide induces shedding of endothelial glycocalyx in coronary vascular bed of guinea pig hearts. Am J Physiol Heart Circ Physiol. 2005 Nov;289(5):H1993-9. doi: 10.1152/ajpheart.00218.2005. Epub 2005 Jun 17. PMID 15964925
- [Background] Bruegger D, Schwartz L, Chappell D, Jacob M, Rehm M, Vogeser M, Christ F, Reichart B, Becker BF. Release of atrial natriuretic peptide precedes shedding of the endothelial glycocalyx equally in patients undergoing on- and off-pump coronary artery bypass surgery. Basic Res Cardiol. 2011 Nov;106(6):1111-21. doi: 10.1007/s00395-011-0203-y. Epub 2011 Jul 19. PMID 21769675
- [Background] Alphonsus CS, Rodseth RN. The endothelial glycocalyx: a review of the vascular barrier. Anaesthesia. 2014 Jul;69(7):777-84. doi: 10.1111/anae.12661. Epub 2014 Apr 28. PMID 24773303
- [Background] Bark BP, Persson J, Grande PO. Importance of the infusion rate for the plasma expanding effect of 5% albumin, 6% HES 130/0.4, 4% gelatin, and 0.9% NaCl in the septic rat. Crit Care Med. 2013 Mar;41(3):857-66. doi: 10.1097/CCM.0b013e318274157e. PMID 23318490
- [Background] Micek ST, McEvoy C, McKenzie M, Hampton N, Doherty JA, Kollef MH. Fluid balance and cardiac function in septic shock as predictors of hospital mortality. Crit Care. 2013 Oct 20;17(5):R246. doi: 10.1186/cc13072. PMID 24138869
- [Background] Boyd JH, Forbes J, Nakada TA, Walley KR, Russell JA. Fluid resuscitation in septic shock: a positive fluid balance and elevated central venous pressure are associated with increased mortality. Crit Care Med. 2011 Feb;39(2):259-65. doi: 10.1097/CCM.0b013e3181feeb15. PMID 20975548
- [Background] Kelm DJ, Perrin JT, Cartin-Ceba R, Gajic O, Schenck L, Kennedy CC. Fluid overload in patients with severe sepsis and septic shock treated with early goal-directed therapy is associated with increased acute need for fluid-related medical interventions and hospital death. Shock. 2015 Jan;43(1):68-73. doi: 10.1097/SHK.0000000000000268. PMID 25247784
- [Background] Maitland K, Kiguli S, Opoka RO, Engoru C, Olupot-Olupot P, Akech SO, Nyeko R, Mtove G, Reyburn H, Lang T, Brent B, Evans JA, Tibenderana JK, Crawley J, Russell EC, Levin M, Babiker AG, Gibb DM; FEAST Trial Group. Mortality after fluid bolus in African children with severe infection. N Engl J Med. 2011 Jun 30;364(26):2483-95. doi: 10.1056/NEJMoa1101549. Epub 2011 May 26. PMID 21615299
- [Background] Kaukonen KM, Bailey M, Pilcher D, Cooper DJ, Bellomo R. Systemic inflammatory response syndrome criteria in defining severe sepsis. N Engl J Med. 2015 Apr 23;372(17):1629-38. doi: 10.1056/NEJMoa1415236. Epub 2015 Mar 17. PMID 25776936
- [Background] Heyland DK, Muscedere J, Drover J, Jiang X, Day AG; Canadian Critical Care Trials Group. Persistent organ dysfunction plus death: a novel, composite outcome measure for critical care trials. Crit Care. 2011;15(2):R98. doi: 10.1186/cc10110. Epub 2011 Mar 18. PMID 21418560